CLINICAL TRIAL: NCT03552133
Title: Feasibility of a Variable Carbon Dioxide (CO2) Rebreathe Device ("Smart CO2") to Treat Obstructive Sleep Apnea
Brief Title: Variable Dead Space Rebreathing Device to Treat Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2016-0475; A538500 (Other: UW Madison); SMPH/POP HEALTH SCI/POP HEALTH (Other: UW Madison); 1R21HL137874-01 (NIH)
Record Dates: First submitted 2018-05-07; First posted 2018-06-11 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-10

CONDITIONS: Sleep Apnea, Obstructive; Sleep Apnea, Central
Keywords: variable deadspace; rebreathe; hypercapnic side-effects
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea, Central

STUDY DESIGN:
Intervention Model Description: One control study night vs. two intervention study nights (subject serves as own control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Smart CO2 (Experimental): Effects of rebreathe device over two sleep nights on sleep apnea, hypoxemia, sleep state, and blood pressure.
  Interventions: Device: Smart CO2
- No intervention (No Intervention): Effects of control night, i.e. no intervention on sleep apnea, hypoxemia, sleep state, and blood pressure.

INTERVENTIONS:
Device: Smart CO2 — A lightweight, cylindrical reservoir attached to a face mask which monitors breathing breath-by-breath and automatically adjusts the level of dead space rebreathe volume so that CO2 will be increased and sleep apnea treated.
  Arms: Smart CO2

SUMMARY:
The purpose of this pilot study is to determine the feasibility of using a novel treatment for sleep apnea in which the patient's own exhaled CO2 is tightly controlled and used in a rebreathe system to reduce sleep disordered breathing.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) needs to be treated with devices that will be utilized with greater compliance by patients than is currently the case with positive airway pressure. To this end, the investigators recently showed that increased inspired CO2 via rebreathing was effective in reducing most obstructive and central apneas in OSA patients. Then, the investigator's University of Wisconsin (UW) team of bioengineers, physiologists, and sleep physicians built a novel variable dead space rebreathe device-with no added positive pressure-which monitors breath by breath ventilation and automatically adjusts the rebreathe dead space volume to add or subtract the level of inspired CO2 depending on the degree of sleep disordered breathing. This approach provides the minimum effective CO2 dose needed in individual OSA patients to stabilize central respiratory motor output and to recruit upper airway dilator muscles, thereby treating obstructive and central apneas. The investigators propose to determine the effectiveness of this "Smart CO2" treatment as well as its effects on sleep state stability, sleep quality, and blood pressure in 10 moderate to severe OSA patients studied over several nights. The investigators expect the findings from the proposed study to be sufficient to determine if the "Smart CO2" treatment is a viable approach to OSA treatment worthy of testing in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, inclusive
2. Moderate to severe OSA (Apnea hypopnea index [AHI] >15 events/hr of sleep)
3. Newly diagnosed OSA, or have either refused to or have not tolerated PAP treatment, or are currently using Positive Airway Pressure (PAP) and are willing to hold it during the night of sleep study visits.
4. Willing and able to provide consent to 5 laboratory visits with 4 full nights of sleep study.
5. Self report of still having sleep apnea since the last sleep test (if diagnosis was greater than a year prior).

Exclusion Criteria:

1. BMI >45 kg/m2
2. AHI<15 events/hour on the first night of sleep testing in our research laboratory (Visit 2)
3. Cigarette smoking of 1 pack per day or more within 6 months of screening;
4. Diagnosed heart failure or coronary artery disease.
5. Diagnosed cerebrovascular disease, Transient Ischemic Attack (TIA) or stroke.
6. Diagnosed asthma or chronic obstructive pulmonary disease with significant airways obstruction (FEVI/Forced Vital Capacity <65%)
7. End-stage hepatic or renal disease
8. Significant daytime sleepiness in subjects who have risky occupations or life-style (for example, working in the transportation industry, history of motor vehicle crash, occupation that requires vigilance for safety or performance)
9. Pregnancy (assessed on urine test at V1 in females with childbearing potential)
10. Clinically significant arrhythmia/dysrhythmias on the clinical diagnostic polysomnography (per medical record) or on research polysomnography conducted at V2
11. Established diagnosis of neuromuscular disease (e.g., Parkinsonism, multiple sclerosis, syringomyelia, transverse myelitis, amyotrophic lateral sclerosis, poliomyelitis, Eaton-Lambert, Guillain-Barre, myasthenia gravis, myotonic dystrophy, mononeuritis multiplex, in the setting of polymyositis/dermatomyositis or severe cervical spine disease)
12. Any current use of benzodiazepines, opioids, or barbiturates
13. Any medical or psychiatric condition which in the opinion of the medical director interferes with the subject's ability to enroll or to continue in the study (once enrolled)
14. Veteran, cared for in the VA system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08; Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Aim 1: Determine the effects of Smart CO2 Device on AHI | three to six weeks
  To determine the effects of a novel, adjustable CO2 rebreathing device on the occurrence of sleep apnea (AHI) in patients with moderate to severe obstructive sleep apnea.
Determine the effect of Smart C02 Device on Arousal Index | three to six weeks
  To determine the effects of a novel, adjustable CO2 rebreathing device on the occurrence of sleep apnea (Arousal Index) in patients with moderate to severe obstructive sleep apnea.

SECONDARY OUTCOMES:
Aim 2: Effect on Sleep state stability | Three to six weeks
  To determine whether this novel treatment influences sleep state stability following sleep.
Determine the effects of Smart CO2 device on Blood pressure (both systolic and diastolic measures) | Three to six weeks
  To determine whether this novel treatment influences systolic or diastolic blood pressure following sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A Dempsey, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No